CLINICAL TRIAL: NCT01129310
Title: A Multicentre, Open-label Phase II Study of Irinotecan, Capecitabine(Xeloda), and Oxaliplatin (IXO) as First Line Treatment in Patients With Metastatic Gastric or Gastroesophageal (GEJ) Adenocarcinoma.
Brief Title: First Line Study of Irinotecan, Capecitabine and Oxaliplatin in Metastatic Gastric or Gastroesophageal Cancer.
Acronym: IXOGoo1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IXOGoo1 25412
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2016-01

CONDITIONS: Gastrointestinal Neoplasm; Gastric Adenocarcinoma
Keywords: irinotecan; capecitabine; oxaliplatin; health-related quality of life; gastroesophageal(GE) junction adenocarcinoma
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Irinotecan; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Irinotecan-Capecitabine-Oxaliplatin — Irinotecan-160mg/m2 IV infusion over 60-90 min on Day 1 Capecitabine-1900mg/m2 daily PO in divided doses (=950mg/m2 BID) on days 2-15 Oxaliplatin- 100mg/m2 IV infusion over 2 hours Day 1
  Other Names: Camptosar; Xeloda; Eloxatin

SUMMARY:
The investigators hypothesize IXO chemotherapy will have an improvement in response rate and acceptable toxicity for uncurable metastatic gastric cancer compared to historical controls.

DETAILED DESCRIPTION:
This is a single arm, open-label, multicentre, phase II trial in which patients with metastatic gastric or GEJ adenocarcinoma will be treated with the combination of irinotecan, capecitabine, and oxaliplatin (IXO).Patients will receive the combination of irinotecan, capecitabine, and oxaliplatin at the recommended phase II dose and sequence determined by the completed phase I trial. Patients will be treated on study until disease progression, overwhelming toxicity, or consent withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* histologically documented gastric GEJ adenocarcinoma not previously treated with palliative systemic therapy.
* Metastatic disease based on the presence of clinically and/or radiologically documented measurable disease based on RECIST.
* ECOG performance status of 0,1 or 2.
* Age ≥ 18 years
* Life expectancy of least 3 months based on discretion of treating oncologist.
* Adequate hematologic, hepatic, and renal function.
* Patients who have received prior chemotherapy or radiation delivered as part of initial curative therapy (i.e. neoadjuvant or adjuvant chemotherapy administered alone and/or concurrently delivered with radiation and/or surgery) are permitted as long as that treatment was completed at least 6 months prior to study start date.
* Patients may have received prior palliative radiotherapy (unless radiation was curative therapy to pelvis or to ≥25% of bone marrow stores) if this radiation was ≥ 4 weeks before study entry and patients must have recovered from the toxic effects of this treatment.
* Patients may have received prior surgery if this surgery was ≥ 4 weeks before study entry and patients must have recovered from the toxic effects of this treatment.
* Patients must have the ability to read, understand, and sign an informed consent and must be willing to comply with study treatment and follow-up.

Exclusion Criteria:

* Patients who have received palliative chemotherapy for their metastatic gastric or GEJ tumor.
* Prior treatment with > 6 cycles of traditional alkylating agent-based chemotherapy, > 2 cycles of carboplatin-based chemotherapy, prior treatment with irinotecan or oxaliplatin chemotherapy, or concurrent treatment with other experimental drugs or anti-cancer therapy.
* Curative radiation treatment to the pelvis or radiation therapy to ≥ 25% of bone marrow stores.
* Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, short gut syndrome, or history of bowel obstruction due to peritoneal metastases.
* Previous of concurrent malignancies, excluding curatively treated in situ carcinoma of the cervix or non-melanoma skin cancer, unless at least 5 years have elapsed since last treatment and the patient is considered cured.
* Any serious medical condition within 6 months prior to study entry such as myocardial infarction, uncontrolled congestive heart failure,unstable angina, active cardiomyopathy, unstable ventricular arrhythmia, cerebrovascular diseases, uncontrolled hypertension, uncontrolled diabetes, uncontrolled psychiatric disorder, serious infection, active peptic ulcer disease, or other medical condition that .....
* Gilbert's disease
* Known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Pre-existing neuropathy ≥ grade 2 from any cause.
* Patients with unstable metastasis to the central nervous system are excluded. Patients who have treated brain metastasis and are off steroids, anticonvulsants, and have documented stability of lesions for at least 3 months may be eligible. A CT scan or MRI is NOT required to rule out brain metastases unless there is clinical suspicion of CNS involvement.
* Pregnant of lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-07; Primary Completion 2018-05-18 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate and dose limiting toxicity | 2 years

SECONDARY OUTCOMES:
Progression Free Survival, overall survival, death, alterations in quality of life outcomes | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Spratlin, MD, Study Chair — Alberta Health services
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada